CLINICAL TRIAL: NCT07368959
Title: ASTRA: A Phase 3 Multi-center, Randomized, Double-Masked, Prospective Study of AURN001 in Subjects With Corneal Edema Secondary to Corneal Endothelial Dysfunction (ABA-3)
Brief Title: AURN001 Efficacy in Participants With Corneal Edema Secondary to Corneal Endothelial Dysfunction
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Aurion Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABA-3
Record Dates: First submitted 2026-01-23; First posted 2026-01-27 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Corneal Edema; Corneal Endothelial Dysfunction; Fuchs Endothelial Corneal Dysfunction; Pseudophakic Bullous Keratopathy (PBK)
Keywords: Best Corrected Visual Acuity; Central corneal thickness; Human Corneal Endothelial Cells; Neltependocel; Postsurgical endothelial dysfunction; Keratoplasty; Pseudophakic Corneal Edema (PCE); Corneal Endothelial Cells; Endothelial Cells; AURN001; Y-27632; Endothelial Keratoplasty; Corneal Endothelial Cell Therapy
MeSH Terms: conditions — Corneal Edema | interventions — Y 27632

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AURN001 (Experimental): Participants will receive single dose of AURN001
  Interventions: Drug: Combination Product: AURN001 + Y-27632
- Placebo (Placebo Comparator): Participants will receive single dose of placebo control.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Combination Product: AURN001 + Y-27632 — AURN001 will be injected to the anterior chamber of the eye.
  Arms: AURN001
Other: Placebo — Placebo control will be injected to the anterior chamber of the eye.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of single injection dose of AURN001 compared with placebo in adult participants with corneal edema secondary to corneal endothelial dysfunction.

ELIGIBILITY:
Key Ocular Inclusion Criteria:

(All ocular criteria apply to the study eye unless noted otherwise)

* Have corneal edema secondary to corneal endothelial dysfunction, requiring surgery (full- or partial-thickness endothelial keratoplasty)
* BCVA between 65 ETDRS letters (approximate 20/50 Snellen equivalent) and 5 ETDRS letters (approximate 20/800 Snellen equivalent)
* Be pseudophakic with PCIOL

Key Ocular Exclusion Criteria:

(All ocular criteria apply to the study eye unless noted otherwise)

* Have progressive corneal dystrophies or degenerations
* Have visually significant corneal or other ocular pathologies

Other inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who achieve a ≥ 15-letter improvement (3-line gain) from baseline in Best Corrected Visual Acuity (BCVA) at Month 6 | At Month 6

SECONDARY OUTCOMES:
Change from baseline in non-contact Central Corneal Thickness (CCT) at Month 6 | Baseline (Day 1) and At Month 6
Change from baseline in BCVA at Month 6 | Baseline (Day 1) and At Month 6

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Investigational Site 2, Mesa, Arizona
  - Investigational Site 6, Little Rock, Arkansas
  - Investigational Site 9, Fort Collins, Colorado
  - Investigational Site 7, Atlanta, Georgia
  - Investigational Site 4, Kansas City, Missouri
  - Investigational Site 11, Leland, North Carolina
  - Investigational Site 5, Winston-Salem, North Carolina
  - Investigational Site 3, Cynwyd, Pennsylvania
  - Investigational Site 10, Plymouth Meeting, Pennsylvania
  - Investigational Site 12, Ladson, South Carolina
  - Investigational Site 8, San Antonio, Texas
  - Investigational Site 1, Spring, Texas

IPD SHARING:
Plan to Share IPD: No